CLINICAL TRIAL: NCT01799837
Title: Kinetic Modeling of Norepinephrine Transporter Availability in PTSD
Brief Title: Norepinephrine Transporter Availability in PTSD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Jonathon Nye, Assistant Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00057641; URC-00025435 (Other: Other)
Record Dates: First submitted 2012-12-13; First posted 2013-02-27 (Estimated); Last update posted 2013-09-11 (Estimated); Status verified 2013-09

CONDITIONS: Posttraumatic Stress Disorder
Keywords: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

ARMS (2):
- Healthy Controls (Other): Posttraumatic stress disorder (PTSD) is a potentially debilitating anxiety disorder triggered when a person is exposed to a traumatic event that is beyond what is experienced in everyday life. A traumatic event may include an interpersonal event like physical or sexual assault, exposure to a disaster or accidents, combat or witnessing a traumatic event. Some symptoms of PTSD include not being able to sleep, nightmares, flashbacks of the event and having problems with memory or not being able to focus. You are being asked to volunteer because you are either 1) a normal healthy volunteer or 2) a deployed veteran or non-deployed veteran who is diagnosed with PTSD. We anticipate enrolling 16 subjects; 8 veterans with PTSD and 8 healthy volunteers without PTSD.
  Interventions: Drug: [C-11]MENET
- Veterans with PTSD (Other): Posttraumatic stress disorder (PTSD) is a potentially debilitating anxiety disorder triggered when a person is exposed to a traumatic event that is beyond what is experienced in everyday life. A traumatic event may include an interpersonal event like physical or sexual assault, exposure to a disaster or accidents, combat or witnessing a traumatic event. Some symptoms of PTSD include not being able to sleep, nightmares, flashbacks of the event and having problems with memory or not being able to focus. You are being asked to volunteer because you are either 1) a normal healthy volunteer or 2) a deployed veteran or non-deployed veteran who is diagnosed with PTSD. We anticipate enrolling 16 subjects; 8 veterans with PTSD and 8 healthy volunteers without PTSD.
  Interventions: Drug: [C-11]MENET

INTERVENTIONS:
Drug: [C-11]MENET — PET imaging involves injecting small amounts of a radioactive material into the blood stream. The radioactive material is attached to a drug called MENET that will give information about how the brain interacts with a protein called norepinephrine (NE).
  Other Names: (2S,3S)-2-[alpha-(2-[11C]- methylphenoxy)phenylmethyl]morpholine([11C]MENET)

SUMMARY:
The objective of this proposal is to collect pilot data to characterize the binding of [11C]MENET in combat-exposed war veterans with posttraumatic stress disorder (PTSD). Approximately two hundred thousand veterans will be returning stateside upon the end of combat operations in Iraq, and 13% of returning veterans will have PTSD. 15% of all war veterans will develop chronic PTSD symptoms requiring a lifetime of mental health care. Little is known about the dysregulation of PTSD veteran's neurochemical state including the noradrenergic system which plays a primary role in memory and stress response. This includes heightened anxiety, fear and hyperarousal symptoms characteristic of PTSD. The noradrenergic system is a concentration of neurons in the brainstem nucleus, locus coerulues, that have projections to the amygdale and prefrontal cortex. The norepinephrine transporter (NET) is responsible for regulating and terminating noradrenergic transmission, and is a specific marker for neuronal integrity. Hyperactivity of the noradrenergic system up-regulates NET protein. An unresolved problem in studying the noradrenergic system is identification of suitable radiopharmaceutical to non-invasively measure alterations in the density of NET. The investigators propose to address this challenge by using positron emission tomography (PET) to measure stress-induced changes in NET expression in combat-exposed war veterans with PTSD. The central hypothesis of this proposal is that war veterans with PTSD have an up-regulation of NET in the locus coerulues resulting from hyperactivity of the noradrenergic system compared to healthy controls. Through a series of experiments, the investigators will determine the in vivo binding characteristics of [11C]MENET. The investigators will use this information to optimally design an experimental protocol to measure the availability of NET in a pilot group of combat-exposed war veterans with PTSD. The aims of this proposal are: 1) Measure the uptake kinetics and whole brain distribution of [11C]MENET in combat-exposed veterans with PTSD and healthy controls, 2) Develop a quantitative kinetic model of [11C]MENET uptake to calculate the NET availability in brain. The subjects undergoing imaging in this work will be recruited by Dr. J. Douglas Bremner (Co-Investigator) at Emory University and Atlanta Veteran Affairs Hospital. Our long-term goal is to develop a longitudinal study framework to assess the NETs dysregulation during onset of PTSD as well as its transition to chronic lifetime PTSD.

ELIGIBILITY:
Inclusion Criteria:

* PTSD as determined by the Structural Clinical Interview for DSMIV (SCID) interview of PTSD and the Clinical Administered PTSD Scale (CAPS).
* Veteran with history of active duty service and currently discharged from active duty service
* Free of psychotropic medication for four weeks before the study

Exclusion Criteria:

* History of shrapnel or other foreign bodies which would preclude MRI scanning
* Meningitis
* Traumatic brain injury
* Neurological disorder or organic mental disorder
* History of loss of consciousness
* Current or lifetime history of alcohol abuse or substance abuse or dependence base on the SCID
* Current or lifetime history of schizophrenia, schizoaffective disorder, or bulimia based on the SCID
* History of serious medical or neurological illness, such as cardiovascular, gastrointestinal, hepatic, renal, neurologic or other systemic illness
* Evidence of a major or neurological illness on physical examination or as a result of laboratory studies
* positive urine toxicology screen
* Current steroid use

Ages: 30 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-06; Primary Completion 2013-04 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Measurement of norepinephrine availability | Participants will be followed for the duration of the hospital stay, an expected average of 1 day
  Information to be obtained are [11C]MENET PET scans including arterial blood sampling to measure blood metabolites.[11C]MENET PET images will be analyze with a full compartmental kinetic analysis. Arterial blood and reference tissue input functions will be used to calculate the distribution volume ratio and binding potential of NET availability in each group

CONTACTS AND LOCATIONS:
Overall Officials: Jonathon A Nye, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States